CLINICAL TRIAL: NCT00702871
Title: A Clinico-Bacteriological Study and Effect of Stress Ulcer Prophylaxis on Occurrence of Ventilator Associated Pneumonia: a Randomized Prospective Study
Brief Title: A Clinico-Bacteriological Study and Effect of Stress Ulcer Prophylaxis on Occurrence of Ventilator Associated Pneumonia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Maulana Azad Medical College (Other)
Responsible Party: Dr Mradul K Daga, Maulana Azad Medical College and Lok Nayak Hospital, Delhi, India
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 403(7)/04MC(ACA)/Protocol/3499
Record Dates: First submitted 2008-06-19; First posted 2008-06-20 (Estimated); Last update posted 2008-06-20 (Estimated); Status verified 2008-06

CONDITIONS: Ventilator Associated Pneumonia; Etiological Organisms; Antimicrobial Drug Susceptibility Pattern; Stress Ulcer Prophylaxis
Keywords: Ventilator Associated Pneumonia; antimicrobial susceptibility pattern; stress ulcer prophylaxis
MeSH Terms: conditions — Pneumonia, Ventilator-Associated | interventions — Ranitidine; Sucralfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Arm 1 was given Injection Ranitidine 50mg i.v. 8 hourly for stress ulcer prophylaxis.
  Interventions: Drug: Ranitidine
- 2 (Active Comparator): In arm 2, Sucralfate was given in dose of 1gm via nasogastric tube 6 hourly for entire duration of ICU stay
  Interventions: Drug: Sucralfate

INTERVENTIONS:
Drug: Ranitidine — In arm 1 Ranitidine was given in dose of 50mg i.v. 8 hourly for entire duration of ICU stay.
  Arms: 1
Drug: Sucralfate — In arm 2, Sucralfate was given in dose of 1gm via nasogastric tube 6 hourly for entire duration of ICU stay
  Arms: 2

SUMMARY:
Objective of this study was to determine incidence, risk factors, etiological micro-organisms and their antimicrobial susceptibility pattern and outcome of VAP; and to study effect of ranitidine vs. sucralfate, used for stress ulcer prophylaxis, on gastric colonization and on occurrence of VAP.

Methods: Design: Prospective randomized study. Setting: ICUs of Medicine Department and Anesthesiology Department, Maulana Azad Medical College and Lok Nayak Hospital, University of Delhi, New Delhi. Patients: 50 patients of age more than 12 years, who had been on ventilator for more than 48 hrs. Intervention: Endotracheal Aspirate and blood sample of all patients were cultured to determine micro-organisms causing VAP and their antimicrobial susceptibility pattern. Patients were divided into 2 groups on random basis. The first group was given ranitidine for stress ulcer prophylaxis while the second was given sucralfate. Thereafter, difference in gastric colonization (on basis of quantitative culture of nasogastric aspirate) and on occurrence of VAP in both the groups was compared.

Study Hypothesis: Study was designed to create data about Ventilator associated pneumonia in developing countries like India. This data is crucial for providing information for deciding future guidelines for treatment of and prevention of Ventilator associated pneumonia. Further to test the hypothesis that H2 blockers, by virtue of raising gastric Ph, increase gastric colonization by pathogenic organism and increase incidence of Ventilator associated pneumonia; patients were divided into two groups on random basis, as described above.

DETAILED DESCRIPTION:
Study population: Fifty patients of either sex admitted to Medical Intensive Care Unit and Intensive Care Unit of Anaesthesiology department of Maulana Azad Medical College and Lok Nayak Hospital, New Delhi( a 2000 bedded, tertiary care centre), fulfilling the criteria were enrolled and prospectively followed up until one week after discharge from intensive care unit or till death.

Methodology: Ventilator associated pneumonia was diagnosed when new and persistent pulmonary infiltrates (not otherwise explained) appeared on chest radiograph after 48 hours of ventilation and any two of the following three criteria were fulfilled:

1. Temperature of more than 38oC or less than 35oC.
2. Leukocytosis ≥16,000 or leukopenia ≤ 3,000.
3. Purulent endotracheal aspirate and/or positive endotracheal aspirate culture. Protocol of study: All patients were ventilated by orotracheal or tracheostomy tube, which was changed only if, blocked or displaced. Patients were ventilated in supine position with frequent changing to right lateral and left lateral positions and nasogastric tube was put in all patients. No prophylactic topical oropharyngeal antibiotic and selective gut decontamination was done in any of the patients. Base line complete blood count was done in all patients at time of intubation. Subsequent counts were done when pneumonia was suspected by onset of fever, new chest signs, worsening of ventilatory requirement and radiologically new infiltrates. Baseline chest X-ray and endotracheal aspirate culture was done at intubation and at 48 hours of ventilation and subsequently done at suspicion of pneumonia or any other pulmonary complications, 48 hours after pneumonia has been detected, routinely once a week if no pneumonia is detected. Nasogastric aspirate culture was done on 3rd and 7th day of intubation and every week thereafter. Gastric colonization was diagnosed if more than 103 colony-forming units/ml were found. Clinical examination for pneumonia and chest radiographs after one week of extubation were done on follow up.

Method of collection of samples: Endotracheal aspirate was collected with mucus trap under all aseptic precautions. Nasogastric (NG) aspirate was collected from indwelling NG tubes. After removing the initial 5 ml, the next 10 ml of fluid in the tube was aspirated into a sterile syringe and immediately transported to the laboratory for processing.

Culture method: A Semi quantitative culture of the endotracheal aspirate and nasogastric aspirate was done [6]. A Measured amount of aspirate was plated on blood agar and Mac-Conkey medium and a colony count was done after incubation. A sample of blood was collected in glucose broth and after overnight incubation, subcultures were done on blood agar and Mac-Conkey agar. Colony characteristics were observed and identification was done in accordance with standard recommendations. Susceptibility of the organisms isolated from endotracheal aspirate was done by disc diffusion technique employing the Stokes method.

Grouping of patients: Patients enrolled into study were divided randomly into two groups on random basis. One group was given Ranitidine (H2 blocker) 50 mg I.V. every 8 hourly as stress ulcer prophylaxis while the other group recieved Sucralfate (surface active agent) 1g 6 hourly via nasogastric tube. Occurrence of VAP in each group was recorded and compared. Gastric colonization in each group was monitored by semi-quantitative culture.

Risk factors studied were age, sex, underlying disease, prior respiratory disease including Chronic obstructive airway disease (COPD), prior hospitalization, duration of intubation, numbers of intubations, prior antibiotic therapy etc. Other parameters noted were indication of mechanical ventilation and outcome of patients with VAP Statistical methods: Incidence, risk factors, outcome and antimicrobial susceptibility were calculated in absolute numbers and percentages. Comparison of effect of ranitidine vs. sucralfate on occurrence of VAP was done by chi square test and effect of ranitidine vs. sucralfate on gastric colonization was calculated in absolute numbers and percentages and compared. All statistics were calculated using SPSS software. P value <0.05 was considered significant.

RISK FACTORS studied include age, sex, underlying disease, prior COPD, prior hospitalization, duration of intubation, no. of intubation. Longer duration of dependence on ventilator increased the risk for VAP significantly (p value 0.001). Similarly, reintubation also emerged as clear predisposing factor for VAP (See table 1).

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 12 years
* Those on mechanical ventilation for more than 48 hours.

Exclusion Criteria:

* Pre-existing pneumonia at the beginning of ventilation or
* Developing pneumonia within 48 hours of ventilation.
* Patients on oral antibiotics

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2005-03; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Occurence of ventilator associated pneumonia | till discharge from ICU or death of Patient

CONTACTS AND LOCATIONS:
Overall Officials: Rajiv Singla, M.D., Principal Investigator — Maulana Azad Medical College and Lok Nayak Hospital, Delhi, India
Locations (1):
- Maulana Azad Medical College and Lok Nayak Hospital, Delhi, National Capital Territory of Delhi, India